CLINICAL TRIAL: NCT05854888
Title: Perineal Massage and Warm Compresses During Second Stage of Labor - Randomised Controlled Trial for Reduce Perineal Trauma
Brief Title: Perineal Massage and Warm Compresses - RCT for Reduce Perineal Trauma During Labor
Acronym: PeMWaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Sílvia Leite Rodrigues, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201802476
Record Dates: First submitted 2023-04-23; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Perineal Tear Resulting From Childbirth
Keywords: Perineum
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The present study was a single-centre, prospective, randomized controlled trial. Eligibility and informed consent to participate were checked once the woman was in established labor. All participants signed an informed consent form and received a copy wherein the study was described in detail.Eligible participants were randomized at the second stage of labor.The trial intervention took place during the second stage of the spontaneous vaginal birth. Participants were randomized to one of the two groups, perineal massage and warm compresses on second stage of labor or control group (hands-on). The participants could adopt the birth position they preferred.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization envelope was opened by the midwife when the participant entered the second stage of labor and was destroyed thereafter. The allocation was only shown to the midwife and if necessary, the obstetrician. The trial intervention took place during the second stage of the spontaneous vaginal birth. Participants were randomized to one of the two groups, perineal massage and warm compresses on second stage of labor or control group (hands-on). The participants were blinded to their allocation. After the placenta delivery, a blinded midwife not otherwise involved in the birth but trained, assessed the perineum (graded the perineal tears). The data about the variables included in the study were registered by the midwife responsible for the birth. Midwives who assess the primary outcomes and the principal investigator were blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeMWaC (Perineal Massage and Warm Compresses) (Experimental): In the second stage of labor, the midwife performed a soft perineal massage between 3 o'clock and 9 o'clock positions (U-shaped reciprocating motion) wearing sterile gloves and lubricated their hand with sterile lubricant. The massage lasted 10 minutes and the degree of downward pressure by the thumb was determined according to mothers' response. Perineal massage was established on the II Hodge Plan, between maternal contractions and regardless of maternal position. The women could adopted the birthing position they prefer. The application of warm compresses was performed by the midwife between the III and IV Hodge plans, during pushing and regardless of the mother's position. A metal jug filled with warm water (between 45° and 59°C) was used to soak the compresses, which were squeezed out before being gently placed on the perineum during contractions.
  Interventions: Procedure: Perineal Massage and Warm Compresses (PeMWaC)
- Control group (Hands-on) (Active Comparator): The midwife placed the index, middle, and little fingers of the non-dominant hand together on the child's occiput, with the palm facing the anterior region of the perineum, when the child's head was crowning. In this way, the expulsion was controlled, maintaining the flexion of the head. Simultaneously, the dominant hand was flattened and placed on the posterior region of the perineum, with the index finger and thumb, forming a "U", exerting pressure on the posterior region of the perineum during the crowning process. During the birth of the shoulders and the rest of the body, the dominant hand was kept in place, protecting the posterior region of the perineum, while the non-dominant hand supported the infant's head, allowing external rotation and spontaneous birth of the shoulders. After both shoulders were removed, the midwife removed the dominant hand from the posterior perineum.
  Interventions: Procedure: Control Group (Hands-on)

INTERVENTIONS:
Procedure: Perineal Massage and Warm Compresses (PeMWaC) — Perineal Massage was performed in the II Hodge Plan, between maternal contractions and regardless of maternal position. Warm Compresses were applied by the midwife between Hodge plans III and IV, during pushing and regardless of maternal position.
  Arms: PeMWaC (Perineal Massage and Warm Compresses)
Procedure: Control Group (Hands-on) — The midwife placed the index, middle, and little fingers of the non-dominant hand together on the child's occiput, with the palm facing the anterior region of the perineum, when the child's head was crowning. In this way, the expulsion was controlled, maintaining the flexion of the head. Simultaneously, the dominant hand was flattened and placed on the posterior region of the perineum, with the index finger and thumb, forming a "U", exerting pressure on the posterior region of the perineum during the crowning process. During the birth of the shoulders and the rest of the body, the dominant hand was kept in place, protecting the posterior region of the perineum.
  Arms: Control group (Hands-on)

SUMMARY:
The aim of this study is to evaluate the effect of a combined perineal massage and warm compresses intervention on the perineum integrity during second stage of labor.

DETAILED DESCRIPTION:
A single-centre, prospective, randomized controlled trial was conducted. Eligibility and informed consent to participate were checked once the woman was in established labor. Eligible participants were randomized at the second stage of labor. The trial intervention took place during the second stage of the spontaneous vaginal birth. Participants were randomized to one of the two groups, perineal massage and warm compresses on second stage of labor or control group (hands-on).

ELIGIBILITY:
Inclusion Criteria:

* Women with 18 years or older
* Between 37 and 41 weeks of pregnancy
* Expected spontaneous vaginal birth
* Fetus in the cephalic presentation
* Able to provide informed written consent

Exclusion Criteria:

* Multiple pregnancy
* Meconial amniotic fluid
* Fetal distress
* Suspicion of fetal growth restriction
* Gestational hypertensive disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Intact Perineum | up to 10 minutes after childbirth
  Absence of tissue separation at any site, without vaginal tears or any other degree of perineal trauma)
First-degree perineal tear | up to 10 minutes after childbirth
  Skin and vaginal tear
Second-degree perineal tear | up to 10 minutes after childbirth
  Skin and muscle tear (posterior compartment)
OASIS | up to 10 minutes after childbirth
  Obstetric anal sphincter injuries (Third-degree tears (injury of anal sphincter) and Fourth-degree tears (Injury of anal sphincter and the anal canal or rectum) without episiotomy
OASIS + episiotomy | up to 10 minutes after childbirth
  Third and fourth degree tear with episiotomy
Episiotomy | up to 10 minutes after childbirth
  without spontaneous perineal trauma or vaginal tears
Episiotomy and first degree tear | up to 10 minutes after childbirth
  Episiotomy with spontaneous skin tear
Episiotomy and second degree tear | up to 10 minutes after childbirth
  Episiotomy and spontaneous skin and muscle tear
OASIS with/without episiotomy | up to 10 minutes after childbirth
  with and without episiotomy
Vaginal tears | up to 10 minutes after childbirth
  only vaginal tear
Anterior Compartment tears | up to 10 minutes after childbirth
  Without episiotomy or any other degree of perineal trauma

SECONDARY OUTCOMES:
Admission to Neonatal Intensive Unit Care | up to 2 hours after childbirth
  Admission to Neonatal Intensive Unit Care
Apgar 5 minutes | 5 minutes after childbirth
  Apgar Score at 5 minutes (0-10) higher scores mean better outcome
Maternal satisfaction with intervention | 24 hours after childbirth
  Question about maternal satisfaction with intervention
Recommend an intervention allocated to a friend | 24 hours after childbirth
  Question about whether women would recommend the intervention they received to a friend
Female Sexual Function Index score | 24 hours, 3 months and 6 months after childbirth
  Female Sexual Function Index score (2-36) higher scores mean better outcome
Pelvic Floor Dysfunction symptoms | 24 hours, 3 months and 6 months after childbirth
  Pelvic Floor Distress Inventory (0-300) higher scores mean worse outcome
Maternal Pain | 24 hours, 3 months and 6 months after childbirth
  Numerical Pain score (0-10) higher scores mean worse outcome
Breastfeeding | 24 hours, 3 months and 6 months after childbirth
  Exclusive breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Sílvia Rodrigues, PhD, Principal Investigator — Institute Biomedical Sciences Abel Salazar-University of Porto
Locations (1):
- Sílvia Rodrigues, Braga, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: up to 3 years after completed the data collection
Access Criteria: Will be shared with other researchers as long as they are involved in research projects

REFERENCES:
- [Derived] Rodrigues S, Silva P, Borges AC, de Sousa NQ, Silva JN, Escuriet R. Effect of Perineal Massage and Warm Compresses Technique in Postpartum Pelvic Floor Dysfunction. A Secondary Analysis from a Randomised Controlled Trial. Reprod Sci. 2024 Apr;31(4):1006-1016. doi: 10.1007/s43032-023-01424-4. Epub 2023 Dec 14. PMID 38097899